CLINICAL TRIAL: NCT04811495
Title: Effectiveness of a Physiotherapy Treatment for Temporomandibular Hyperlaxity: a Case Report.
Brief Title: Effectiveness of a Physiotherapy Treatment for Temporomandibular Hyperlaxity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Clinical Professor, Universidad Católica de Ávila
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19/03/2021
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Disorders, Temporomandibular Joint; Range of Motion, Articular
Keywords: range of motion, articular; disorders, temporomandibular joint
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with temporomandibular joint disorders (Experimental)
  Interventions: Other: Physiotherapy treatment

INTERVENTIONS:
Other: Physiotherapy treatment — A treatment plan is carried out which aims to improve pain, muscle balance and range of motion of the temporomandibular joint.

SUMMARY:
A 14-day physiotherapy treatment for temporomandibular joint hyperlaxity is established. Pre-intervention measurements and intermediate and end-of-treatment measurements are taken. Range of movement, algometry and muscle balance are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Woman with temporomandicular joint pain for six months and diagnosed with hyperlaxity in the joint.

Exclusion Criteria:

* Men
* No temporomandibular joint pain or hyperlaxity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Range motion | 14 days
  The range of movement in the temporomandibular joint is assessed.
VAS | 14 days
  Pain in the temporomandibular artiuclation measured with an algometer and VAS is assessed.
Strength | 14 days
  The strength of the temporomandibular joint musculature measured with an algometer is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buvinic S, Balanta-Melo J, Kupczik K, Vasquez W, Beato C, Toro-Ibacache V. Muscle-Bone Crosstalk in the Masticatory System: From Biomechanical to Molecular Interactions. Front Endocrinol (Lausanne). 2021 Mar 1;11:606947. doi: 10.3389/fendo.2020.606947. eCollection 2020. PMID 33732211
- [Result] Al-Jewair T, Shibeika D, Ohrbach R. Temporomandibular Disorders and Their Association with Sleep Disorders in Adults: A Systematic Review. J Oral Facial Pain Headache. 2021 Winter;35(1):41-53. doi: 10.11607/ofph.2780. PMID 33730126
- [Result] Kaya DI, Ataoglu H. Botulinum toxin treatment of temporomandibular joint pain in patients with bruxism: A prospective and randomized clinical study. Niger J Clin Pract. 2021 Mar;24(3):412-417. doi: 10.4103/njcp.njcp_251_20. PMID 33723117
- [Result] Angelo DF, Moreira A, Sanz D, Sao Joao R. Hearing changes after temporomandibular joint arthroscopy: a prospective study. Int J Oral Maxillofac Surg. 2021 Nov;50(11):1491-1495. doi: 10.1016/j.ijom.2021.02.013. Epub 2021 Mar 11. PMID 33714614
- [Result] Candido Dos Reis A, Theodoro de Oliveira T, Vidal CL, Borsatto MC, Lima da Costa Valente M. Effect of Auricular Acupuncture on the Reduction of Symptoms Related to Sleep Disorders, Anxiety and Temporomandibular Disorder (TMD). Altern Ther Health Med. 2021 Mar;27(2):22-26. PMID 33711819
- [Result] Asquini G, Rushton A, Pitance L, Heneghan N, Falla D. The effectiveness of manual therapy applied to craniomandibular structures in the treatment of temporomandibular disorders: protocol for a systematic review. Syst Rev. 2021 Mar 8;10(1):70. doi: 10.1186/s13643-021-01623-7. PMID 33685496
- [Result] Memmedova F, Emre U, Yalin OO, Dogan OC. Evaluation of temporomandibular joint disorder in headache patients. Neurol Sci. 2021 Nov;42(11):4503-4509. doi: 10.1007/s10072-021-05119-z. Epub 2021 Feb 18. PMID 33604763
- [Result] Castien RF, Scholten-Peeters GG. Letter to the Editor concerning 'Effects of physical therapy for temporomandibular disorders on headache pain intensity: A systematic review' by van der Meer et al. Musculoskelet Sci Pract. 2021 Jun;53:102324. doi: 10.1016/j.msksp.2021.102324. Epub 2021 Feb 16. No abstract available. PMID 33602632
- [Result] Wu M, Cai J, Yu Y, Hu S, Wang Y, Wu M. Therapeutic Agents for the Treatment of Temporomandibular Joint Disorders: Progress and Perspective. Front Pharmacol. 2021 Jan 29;11:596099. doi: 10.3389/fphar.2020.596099. eCollection 2020. PMID 33584275
- [Result] Peixoto KO, da Silva Bezerra A, Melo RA, de Resende CMBM, de Almeida EO, Barbosa GAS. Short-Term Effect of Scalp Acupuncture on Pain, Sleep Disorders, and Quality of Life in Patients with Temporomandibular Disorders: A A Randomized Clinical Trial. Pain Med. 2021 Apr 20;22(4):905-914. doi: 10.1093/pm/pnab048. PMID 33561277
- [Result] Onoda N, Mikami T, Saito N, Kobayashi T. Evaluation of oral health-related quality of life in patients with temporomandibular disorders. Cranio. 2023 Nov;41(6):486-493. doi: 10.1080/08869634.2021.1883378. Epub 2021 Feb 8. PMID 33554774
- [Result] Nahian A, Mathew Jr J. Osteopathic Manipulative Treatment: Facial Muscle Energy, Direct MFR, and BLT Procedure - for TMJ Dysfunction. 2023 Feb 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564310/ PMID 33231980